CLINICAL TRIAL: NCT05646108
Title: Tubridge Flow Diverter Study For Intracranial Aneurysms: A Post Market Nationwide Multi-center Registry Study In China
Brief Title: Tubridge Flow Diverter Study For Intracranial Aneurysms
Acronym: TRACE-IA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: MicroPort NeuroTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Tubridge-2022-01-A
Record Dates: First submitted 2022-05-29; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Intracranial Aneurysm
Keywords: flow diverter; Intracranial aneurysm; cerebral aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endovascular treatment — Endovascular treatment

SUMMARY:
The scope of this trial is the collection and analysis of the important safety outcomes in the real world, related to the use of the Tubridge flow diverter in the treatment of intracranial aneurysms.

DETAILED DESCRIPTION:
A cerebral aneurysm (also known as an intracranial or intracerebral aneurysm) is a weak or thin spot on a blood vessel in the brain that balloons out and fills and intermixes with parent artery blood. Incidence of intracranial aneurysms varies by country, with reports of prevalence ranging from 5.1 to 19.6 cases per 100,000 persons. The most devastating presentation of an intracranial aneurysm is subarachnoid hemorrhage (SAH). It is estimated that, on average, five percent of the population is afflicted and the incidence of aneurysm rupture (SAH) is between 6 and 9 per 1000 000 individuals .Mortality can approach 50%, with fewer than 60% of survivors returning to independent living.

Invasive treatment of aneurysms began with an open surgical procedure referred to as 'surgical clipping'. This treatment was once considered the gold standard treatment for aneurysms. Traditional surgery requires craniotomy to reach the aneurysm in the brain and place the clip on the neck (opening) of the aneurysm to block the blood flow into the aneurysm. It usually has a higher complication rate and mortality rate. In contrast to the surgery, endovascular treatment via a minimally invasive procedure Endovascular treatment has become the mainstream treatment of intracranial aneurysms, which consists of coiling, stent-assisted coiling, and flow diversion.

Flow diverter is a stent-like device with low-porosity and higher metal coverage would significantly change the direction of the blood flow, reduce the hemodynamic impact on the aneurysmal necks, and further induce intra-saccular thrombogenesis; also, they would serve as scaffolds to promote intima formation, which has a distinct effect on the healing of aneurysmal necks. Meanwhile, due to the pressure gradient between the main trunk and perforators, those perforators would keep patent. The emergence of the flow diverter shows the treatment of the brain aneurysm changed from the concept of aneurysm sac packing to the hemodynamic reconstruction of the parent vessel.

In recent years, commercialized flow diverter represented as pipeline embolization device (Medtronic, Irvine, California, USA) which is braided strands of cobalt chromium and platinum, and Silk Flow Diverter (Balt Extrusion, Montmorency, France) which is braided from nitinol wires. One potential technical concern with different material or design for FD is that of may lead to different flow reduction effects or mechanical properties, which can result in neurologic complications. Tubridge flow diverter is a self-expended stent which is braided of nickel-titanium microfilaments with two platinum-iridium microfilaments through the entire stent. It has been in commercial clinical use in China since April 2018. Here, the investigator conducted a post market, nationwide, multicenter registry research on embolization of intracranial aneurysms with tubridge flow diverter in China, to evaluate the important clinical outcomes in real-world use.

ELIGIBILITY:
Inclusion Criteria:

* 1. received Tubridge flow diverter treatment for intracranial aneurysm after the date of regulatory approval in China

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
The primary end point was the event-free survival rate at 12 months(Plus 0.5 month). | 12 months (Plus 0.5 month)
  defined as the occurrence of morbidity (ispontaneous rupture of the target aneurysm causing subarachnoid hemorrhage or cavernous carotid fistula, intraparenchymal hemorrhage (IPH)(both ipsilateral and contralateral), ischemic stroke, and permanent cranial neuropathy,or death within 12 months(Plus 0.5 month) post-treatment.For the Tubridge flow diverter, this endpoint will be based upon the evaluation of clinical event committee, identification of patients with neurologic clinical events after Tubridge flow diverter treatment, including but not limited: Spontaneous rupture of the target aneurysm, Intraparenchymal hemorrhage, Ischemic stroke, cranial neuropathy.Transient ischemic stroke without clinical adverse events was not included.

SECONDARY OUTCOMES:
The clinical outcome defined by the mRS at 12 months (Plus 0.5 month) after aneurysm treatment. | 12 months (Plus 0.5 month)
  In patients where mRS at 12months were not available, the last available mRS was used instead;
Occurrence of ipsilateral major stroke or neurovascular death in 1 months (Plus 7 days), including but not limited: Spontaneous rupture of the target aneurysm, ipsilateral intraparenchymal hemorrhage, ipsilateral ischemic stroke, cranial neuropathy. | 1 months (Plus 7 days)
The event-free survival rate at 24 months(Plus 0.5 month); | 24 months(Plus 0.5 month)
The event-free survival rate at 36 months(Plus 0.5 month); | 36 months(Plus 0.5 month)
The event-free survival rate at 48 months(Plus 0.5 month); | 48 months(Plus 0.5 month)
Median event-free survival time | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Ph.D, Study Chair — Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided